CLINICAL TRIAL: NCT00933387
Title: A Phase II Study of Neoadjuvant Bio-chemotherapy With Cetuximab, Paclitaxel, and Cisplatin (CPC) Followed by Cetuximab-based Concurrent Bio-radiotherapy in High-risk Locally Advanced Oral Squamous Cell Carcinoma (OSCC)
Brief Title: A Study of Neoadjuvant Bio-C/T Followed by Concurrent Bio-R/T in High-risk Locally Advanced Oral Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: China Medical University Hospital (Other); National Cheng-Kung University Hospital (Other); Chi Mei Medical Hospital (Other); Changhua Christian Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1309; EMR62202-845
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2009-10

CONDITIONS: Oral Cancer
Keywords: oral squamous cell carcinoma; neoadjuvant bio-chemotherapy; concurrent bio-radiotherapy; biomarker
MeSH Terms: conditions — Mouth Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; TP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open label (Experimental): an open-labelled, single-arm
  Interventions: Drug: Cetuximab,Paclitaxel,Cisplatin

INTERVENTIONS:
Drug: Cetuximab,Paclitaxel,Cisplatin — Cetuximab 500 mg/m2 iv infusion (120 min for the 1st infusion, 90 min for the 2nd , and 60 min for the subsequent) Paclitaxel 120 mg/m2 3-hour iv infusion Cisplatin 50 mg/m2 2-hour iv infusion

SUMMARY:
Surgical resection followed by concurrent chemoradiotherapy is considered as the standard of care for locally advanced OSCC (LAOSCC). Although the treatment could provide prompt local control, but it is also associated with high incidence of distant failure. Systemic chemotherapy given either before (neoadjuvant) or after (adjuvant) definitive local treatment has been extensively evaluated to improve the clinical outcome in LAOSCC. Regimens of taxane/cisplatin-based combinations have been shown to improve the treatment outcome of patients with locally advanced head and neck squamous cell carcinoma (HNSCC) in neoadjuvant setting. Recently, cetuximab (Erbitux®), a monoclonal antibody against epidermal growth factor receptor (EGFR), has also been proven to be an efficient agent for advanced and/or refractory HNSCC with acceptable toxicity profiles. In current study, we shall evaluate the feasibility, efficacy and safety of a triplet bio-chemotherapy consisting of cetuximab, paclitaxel, and cisplatin followed by cetuximab-based concurrent bio-radiotherapy (CBRT) in patients with LAOSCC.

DETAILED DESCRIPTION:
Patients with high-risk, locally advanced (TxN2b~3 or T4N0~3, M0) OSCC will be eligible. To detect an interested objective response rate (p1) of 80% versus a non-interested response (p0) rate of 60%, with an α and 1-β of 0.05 and 0.2, respectively (two-sided test), including the estimated dropout rate of 10%, a total of 47 patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. High-risk, locally advanced (TxN2b~3 or unresectable T4, M0) OSCC
2. Histologically confirmed squamous cell carcinoma
3. Performance status: Eastern Cooperative Oncology Group performance status (ECOG) 0-1
4. age 18 years or older, less than 70 years of age
5. Having signed informed consent
6. Measurable disease by CT or MRI
7. Adequate hematologic, hepatic and renal function

Exclusion Criteria:

1. Prior radiotherapy for targeted lesions, chemotherapy, EGFR pathway targeting therapy
2. Prior surgery for cancer except for the purpose of diagnostic biopsy
3. Concomitant active 2nd malignancies or disease-free of malignancies < 3 years before the study except adequately treated in situ cervical cancer, or non-melanoma skin cancer
4. Concomitant anticancer therapies within the past 28 days
5. Severe cardiopulmonary diseases and other systemic disease under poor control
6. Uncontrolled chronic neuropathy
7. Women who are positive of pregnancy, or in breast-feeding
8. Known allergy to any study treatment
9. Legal incapacity
10. Significant disease which, in the investigator's opinion, would exclude the patient from the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the overall response rate after completion of the assigned treatment. | 18 weeks

SECONDARY OUTCOMES:
Secondary endpoints include the response rate after neoadjuvant therapy, progression-free survival, overall survival, biomarker prediction, and toxicity. | >2 years

CONTACTS AND LOCATIONS:
Overall Officials: J Y Chang, M.D., Principal Investigator — National Health Research of Institutes
Locations (1):
- National Health Research of Institutes, Taiwan Cooperative Oncology Group, Tainan, Taiwan